CLINICAL TRIAL: NCT01375842
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of Atezolizumab (MPDL3280A) Administered Intravenously as a Single Agent to Patients With Locally Advanced or Metastatic Solid Tumors or Hematologic Malignancies
Brief Title: A Study of Atezolizumab (an Engineered Anti-Programmed Death-Ligand 1 [PDL1] Antibody) to Evaluate Safety, Tolerability and Pharmacokinetics in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD4989g; 2011-001422-23 (EudraCT Number); GO27831 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Tumors; Hematologic Malignancies
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — atezolizumab

ARMS (9):
- Dose Escalation Cohort: Atezolizumab 0.01 mg/kg (Experimental): Participants will receive intravenous (IV) infusion of atezolizumab 0.01 milligrams per kilogram (mg/kg) every 3 weeks (q3w) until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 0.03 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 0.03 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 0.1 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 0.1 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 0.3 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 0.3 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 1 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 1 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 3 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 3 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 10 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 10 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Dose Escalation Cohort: Atezolizumab 20 mg/kg (Experimental): Participants will receive IV infusion of atezolizumab 20 mg/kg q3w until DLT is reached or up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first.
  Interventions: Drug: Atezolizumab
- Expansion Cohort (Atezolizumab) (Experimental): Participants will receive IV infusion of atezolizumab q3w up to end of study or treatment discontinuation or death or until initiation of another anti cancer therapy, whichever occurs first. The dose which result in total drug exposure less than or equal to (</=) exposures achieved at the MTD or maximum administered dose (MAD), will be selected for expansion cohort.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as IV infusion at eight dose levels (0.01, 0.03, 0.1, 0.3, 1, 3, 10, 20 mg/kg) in dose escalation cohort and at a dose which result in total drug exposure </= exposures achieved at the MTD or MAD, will be selected for expansion cohort.
  Other Names: MPDL3280A

SUMMARY:
This Phase I, multicenter, first-in-human, open-label, dose-escalation study will evaluate the safety, tolerability, and pharmacokinetics of atezolizumab (MPDL3280A) administered as single agent to participants with locally advanced or metastatic solid malignancies or hematologic malignancies. The study will be conducted in two cohorts: Dose-escalation cohort and Expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 16 to 17 years old would be enrolled after consultation with the Medical Monitor
* Histologically or cytologically documented, incurable or metastatic solid tumor or hematologic malignancy that is advanced (non-resectable) or recurrent and progressing since the last anti-tumor therapy and for which no recognized standard curative therapy exists
* Representative tumor specimens in paraffin blocks (preferred) or at least 15 unstained slides, with an associated pathology report
* Adequate hematologic and end organ function
* Measurable disease per RECIST v1.1 for participants with solid malignancies. Disease-specific criteria for participants with prostate cancer, glioblastoma multiforme (GBM), malignant lymphoma, or multiple myeloma
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* For participants who will undergo serial biopsy in dose-escalation cohort, baseline tumor tissue samples should be of core needle biopsies for deep tumor tissue or organs or excisional or punch biopsies for cutaneous or subcutaneous lesions (>/=5 millimeter [mm] in diameter amenable to serial biopsy)

Exclusion Criteria:

* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases
* Known hypersensitivity to pharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History or risk of autoimmune disease (for example, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis)
* History of human immunodeficiency virus (HIV) infection, active hepatitis B (chronic or acute), or hepatitis C infection
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1
* Malignancies other than disease under study within 5 years prior to Cycle 1, Day 1
* Participants with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Day 1 up to Day 21
Maximum Tolerated Dose (MTD) of Atezolizumab | Day 1 up to Day 21
Recommended Phase 2 Dose (RP2D) of Atezolizumab | Baseline up to time of determination of MTD (up to Day 21)
Percentage of Participants With Adverse Events | Baseline up to 90 days after the last dose of study treatment or until initiation of another anti-cancer therapy, whichever occurs first (up to approximately [approx] 7 years [yrs])

SECONDARY OUTCOMES:
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) | Predose(0 hour[hr])on Day 1 of Cycles 1,2,4,8,16,17,20(Cycle length=21 days), every 8 cycles thereafter, at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure(up to approx 7 yrs)
Area Under the Concentration-Time Curve (AUC) of Atezolizumab | Predose (0 hr) on Day 1 of Cycle 1 up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) (Detailed timeframe provided in outcome measure description)
  Dose-Escalation Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 minutes [min]) on Day 1 of Cycles 1-5, 7 (Cycle length=21 days); Days 2, 4, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 8, 10, 12, 14, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) Expansion Cohort: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 min) on Day 1 of Cycles 1-4 (Cycle length=21 days); Days 2, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 2-5, 7, 8, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs)
Maximum Serum Concentration (Cmax) of Atezolizumab | Predose (0 hr) on Day 1 of Cycle 1 up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) (Detailed timeframe provided in outcome measure description)
  Dose-Escalation Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 minutes [min]) on Day 1 of Cycles 1-5, 7 (Cycle length=21 days); Days 2, 4, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 8, 10, 12, 14, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) Expansion Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 min) on Day 1 of Cycles 1-4 (Cycle length=21 days); Days 2, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 2-5, 7, 8, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs)
Minimum Serum Concentration (Cmin) of Atezolizumab | Predose (0 hr) on Day 1 of Cycle 1 up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) (Detailed timeframe provided in outcome measure description)
  Dose-Escalation Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 minutes [min]) on Day 1 of Cycles 1-5, 7 (Cycle length=21 days); Days 2, 4, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 8, 10, 12, 14, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) Expansion Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 min) on Day 1 of Cycles 1-4 (Cycle length=21 days); Days 2, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 2-5, 7, 8, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs)
Clearance (CL) of Atezolizumab | Predose (0 hr) on Day 1 of Cycle 1 up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) (Detailed timeframe provided in outcome measure description)
  Dose-Escalation Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 minutes [min]) on Day 1 of Cycles 1-5, 7 (Cycle length=21 days); Days 2, 4, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 8, 10, 12, 14, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) Expansion Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 min) on Day 1 of Cycles 1-4 (Cycle length=21 days); Days 2, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 2-5, 7, 8, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs)
Volume at Steady State (Vss) of Atezolizumab | Predose (0 hr) on Day 1 of Cycle 1 up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) (Detailed timeframe provided in outcome measure description)
  Dose-Escalation Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 minutes [min]) on Day 1 of Cycles 1-5, 7 (Cycle length=21 days); Days 2, 4, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 8, 10, 12, 14, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs) Expansion Cohorts: Predose (0 hr), 0.5 hr post-infusion (infusion duration=60 min) on Day 1 of Cycles 1-4 (Cycle length=21 days); Days 2, 8, 15 of Cycle 1; predose (0 hr) on Day 1 of Cycles 2-5, 7, 8, 16, 17, 20, every 8 cycles thereafter (up to approx 7 yrs), at treatment discontinuation & then every 30 days for up to 120 days after last dose of study treatment until death/study closure (up to approx 7 yrs)
Percentage of Participants With Best Overall Response, Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From Baseline up to the first occurrence of progression or death, whichever occurs first (up to approx 7 yrs)
Percentage of Participants With Best Overall Response, Assessed by Immune-Related Response Criteria (irRC) | From Baseline up to the first occurrence of progression or death, whichever occurs first (up to approx 7 yrs)
Percentage of Participants With Objective Response (Complete Response [CR] or Partial Response [PR]), Assessed by RECIST v1.1 | From Baseline up to the first occurrence of progression or death, whichever occurs first (up to approx 7 yrs)
Percentage of Participants With Objective Response (CR or PR), Assessed by irRC | From Baseline up to the first occurrence of progression or death, whichever occurs first (up to approx 7 yrs)
Duration of Objective Response, Assessed by RECIST v1.1 | Time from the first occurrence of a documented objective response to the time of relapse or death from any cause (up to approx 7 yrs)
Duration of Objective Response, Assessed by irRC | Time from the first occurrence of a documented objective response to the time of relapse or death from any cause (up to approx 7 yrs)
Progression-Free Survival (PFS), Assessed by RECIST v1.1 | From Baseline up to the first occurrence of progression or death, whichever occurs first (up to approx 7 yrs)
PFS, Assessed by irRC | From Baseline up to the first occurrence of progression or death, whichever occurs first (up to approx 7 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (21):
- United States (16):
  - HonorHealth Research Institute - Pima Center, Scottsdale, Arizona
  - The Angeles Clinic, Los Angeles, California
  - Stanford Univ Medical Center; Dept Central Pharmacy, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Uni of Chicago, Chicago, Illinois
  - Johns Hopkins Univ Med Center, Baltimore, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - Carolina BioOncology Institute; Can Therapy & Res Ctr, Huntersville, North Carolina
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Virginia Oncology Associates, Norfolk, Virginia
- France (3):
  - Centre Leon Berard, Lyon
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Drct, Villejuif
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Barts & London School of Med; Medical Oncology, London, United Kingdom

REFERENCES:
- [Derived] Petrylak DP, Loriot Y, Shaffer DR, Braiteh F, Powderly J, Harshman LC, Conkling P, Delord JP, Gordon M, Kim JW, Sarkar I, Yuen K, Kadel EE 3rd, Mariathasan S, O'Hear C, Narayanan S, Fasso M, Carroll S, Powles T. Safety and Clinical Activity of Atezolizumab in Patients with Metastatic Castration-Resistant Prostate Cancer: A Phase I Study. Clin Cancer Res. 2021 Jun 15;27(12):3360-3369. doi: 10.1158/1078-0432.CCR-20-1981. Epub 2021 Feb 10. PMID 33568344
- [Derived] Shemesh CS, Chan P, Legrand FA, Shames DS, Das Thakur M, Shi J, Bailey L, Vadhavkar S, He X, Zhang W, Bruno R. Pan-cancer population pharmacokinetics and exposure-safety and -efficacy analyses of atezolizumab in patients with high tumor mutational burden. Pharmacol Res Perspect. 2020 Dec;8(6):e00685. doi: 10.1002/prp2.685. PMID 33241650
- [Derived] Chiang AC, Sequist LVD, Gilbert J, Conkling P, Thompson D, Marcoux JP, Gettinger S, Kowanetz M, Molinero L, O'Hear C, Fasso M, Lam S, Gordon MS. Clinical Activity and Safety of Atezolizumab in a Phase 1 Study of Patients With Relapsed/Refractory Small-Cell Lung Cancer. Clin Lung Cancer. 2020 Sep;21(5):455-463.e4. doi: 10.1016/j.cllc.2020.05.008. Epub 2020 May 12. PMID 32586767
- [Derived] Molinero L, Li Y, Chang CW, Maund S, Berg M, Harrison J, Fasso M, O'Hear C, Hegde P, Emens LA. Tumor immune microenvironment and genomic evolution in a patient with metastatic triple negative breast cancer and a complete response to atezolizumab. J Immunother Cancer. 2019 Oct 23;7(1):274. doi: 10.1186/s40425-019-0740-8. PMID 31647026
- [Derived] Morrissey KM, Marchand M, Patel H, Zhang R, Wu B, Phyllis Chan H, Mecke A, Girish S, Jin JY, Winter HR, Bruno R. Alternative dosing regimens for atezolizumab: an example of model-informed drug development in the postmarketing setting. Cancer Chemother Pharmacol. 2019 Dec;84(6):1257-1267. doi: 10.1007/s00280-019-03954-8. Epub 2019 Sep 21. PMID 31542806
- [Derived] Hamid O, Molinero L, Bolen CR, Sosman JA, Munoz-Couselo E, Kluger HM, McDermott DF, Powderly JD, Sarkar I, Ballinger M, Fasso M, O'Hear C, Chen DS, Hegde PS, Hodi FS. Safety, Clinical Activity, and Biological Correlates of Response in Patients with Metastatic Melanoma: Results from a Phase I Trial of Atezolizumab. Clin Cancer Res. 2019 Oct 15;25(20):6061-6072. doi: 10.1158/1078-0432.CCR-18-3488. Epub 2019 Jul 29. PMID 31358540
- [Derived] Liu JF, Gordon M, Veneris J, Braiteh F, Balmanoukian A, Eder JP, Oaknin A, Hamilton E, Wang Y, Sarkar I, Molinero L, Fasso M, O'Hear C, Lin YG, Emens LA. Safety, clinical activity and biomarker assessments of atezolizumab from a Phase I study in advanced/recurrent ovarian and uterine cancers. Gynecol Oncol. 2019 Aug;154(2):314-322. doi: 10.1016/j.ygyno.2019.05.021. Epub 2019 Jun 14. PMID 31204078
- [Derived] Emens LA, Cruz C, Eder JP, Braiteh F, Chung C, Tolaney SM, Kuter I, Nanda R, Cassier PA, Delord JP, Gordon MS, ElGabry E, Chang CW, Sarkar I, Grossman W, O'Hear C, Fasso M, Molinero L, Schmid P. Long-term Clinical Outcomes and Biomarker Analyses of Atezolizumab Therapy for Patients With Metastatic Triple-Negative Breast Cancer: A Phase 1 Study. JAMA Oncol. 2019 Jan 1;5(1):74-82. doi: 10.1001/jamaoncol.2018.4224. PMID 30242306
- [Derived] Colevas AD, Bahleda R, Braiteh F, Balmanoukian A, Brana I, Chau NG, Sarkar I, Molinero L, Grossman W, Kabbinavar F, Fasso M, O'Hear C, Powderly J. Safety and clinical activity of atezolizumab in head and neck cancer: results from a phase I trial. Ann Oncol. 2018 Nov 1;29(11):2247-2253. doi: 10.1093/annonc/mdy411. PMID 30219915
- [Derived] Horn L, Gettinger SN, Gordon MS, Herbst RS, Gandhi L, Felip E, Sequist LV, Spigel DR, Antonia SJ, Balmanoukian A, Cassier PA, Liu B, Kowanetz M, O'Hear C, Fasso M, Grossman W, Sandler A, Soria JC. Safety and clinical activity of atezolizumab monotherapy in metastatic non-small-cell lung cancer: final results from a phase I study. Eur J Cancer. 2018 Sep;101:201-209. doi: 10.1016/j.ejca.2018.06.031. Epub 2018 Aug 1. PMID 30077125
- [Derived] Lukas RV, Rodon J, Becker K, Wong ET, Shih K, Touat M, Fasso M, Osborne S, Molinero L, O'Hear C, Grossman W, Baehring J. Clinical activity and safety of atezolizumab in patients with recurrent glioblastoma. J Neurooncol. 2018 Nov;140(2):317-328. doi: 10.1007/s11060-018-2955-9. Epub 2018 Aug 2. PMID 30073642
- [Derived] Petrylak DP, Powles T, Bellmunt J, Braiteh F, Loriot Y, Morales-Barrera R, Burris HA, Kim JW, Ding B, Kaiser C, Fasso M, O'Hear C, Vogelzang NJ. Atezolizumab (MPDL3280A) Monotherapy for Patients With Metastatic Urothelial Cancer: Long-term Outcomes From a Phase 1 Study. JAMA Oncol. 2018 Apr 1;4(4):537-544. doi: 10.1001/jamaoncol.2017.5440. PMID 29423515
- [Derived] McDermott DF, Sosman JA, Sznol M, Massard C, Gordon MS, Hamid O, Powderly JD, Infante JR, Fasso M, Wang YV, Zou W, Hegde PS, Fine GD, Powles T. Atezolizumab, an Anti-Programmed Death-Ligand 1 Antibody, in Metastatic Renal Cell Carcinoma: Long-Term Safety, Clinical Activity, and Immune Correlates From a Phase Ia Study. J Clin Oncol. 2016 Mar 10;34(8):833-42. doi: 10.1200/JCO.2015.63.7421. Epub 2016 Jan 11. PMID 26755520
- [Derived] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504